CLINICAL TRIAL: NCT06954896
Title: Comparison of Superior Hypogastric Plexus Block and Peritoneal Bupivacaine in Pain Management After Laparoscopic Hysterectomy
Brief Title: Comparison of Superior Hypogastric Plexus Block and Peritoneal Bupivacaine in Pain Management
Status: Completed | Type: Observational
Sponsor: Enes Celik (Other)
Responsible Party: Sponsor-Investigator, Enes Celik, Anesthesiologist, Mardin Artuklu University
Organization: Mardin Artuklu University (Other)
Other Study IDs: ArtukluU-MED-EC-01
Record Dates: First submitted 2025-04-14; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Superior Hypogastric Plexus Block; Intraperitoneal Bupivacaine
Keywords: Hypogastric Plexus; Hysterectomy; Intraperitoneal Injections
MeSH Terms: interventions — Bupivacaine; dexketoprofen trometamol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- intraperitoneal local anaesthetic spray (Group B)
  Interventions: Drug: Intraperitoneal Bupivacaine spray
- intravenous analgesics (Group C)
  Interventions: Drug: Dexketoprofen (KETAVEL 50 mg/2 ml)
- superior hypogastric plexus block (Group S)
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — The superior hypogastric plexus block (SHPB) was performed following uterine removal and closure of the vaginal cuff, but prior to trocar removal from the abdominal cavity. The promontory was identified under laparoscopic visualization. The posterior peritoneum overlying the promontory was gently grasped and elevated with an instrument to create a peritoneal tent. A needle was then inserted at the apex of the tent and advanced approximately 1 cm. At this point, a subperitoneal space was further expanded using a surgical instrument, and 30 ml of 0.25% bupivacaine was injected into the area
  Groups: superior hypogastric plexus block (Group S)
Drug: Dexketoprofen (KETAVEL 50 mg/2 ml) — In cases where the VAS score exceeded 3 in the postoperative period, it was deemed that the patient's analgesia was insufficient, prompting the intravenous administration of 50 mg of dexketoprofen sodium.
  Groups: intravenous analgesics (Group C)
Drug: Intraperitoneal Bupivacaine spray — The peritoneal cavity and abdominal wall were treated with 30 milliliters of 0.25% bupivacaine, with a focus on areas involving the peritoneum in the lower abdominal region.
  Groups: intraperitoneal local anaesthetic spray (Group B)

SUMMARY:
Background: Laparoscopic hysterectomy is one of the most frequently performed major surgeries in nonmalignant gynecological diseases. Effective postoperative analgesia is associated with short hospital stays, early mobilization, reduced costs, and patient satisfaction. Intravenous administration of nonsteroidal anti-inflammatory drugs, paracetamol or opioids; epidural catheter placement; peritoneal local anaesthetic administration; and superior hypogastric plexus block (SHPB) are routinely employed methods for postoperative pain management following laparoscopic hysterectomy.

Methods: The study population comprised patients who underwent laparoscopic hysterectomy with or without oophorectomy for benign indications. A total of 94 patients were included in the study. Thirty patients received a superior hypogastric plexus block, thirty received intraperitoneal local anaesthetic spray, and thirty-four received intravenous analgesics.

Conclusion: In the present study, a comparison of postoperative pain management in patients who underwent laparoscopic hysterectomy was conducted.

DETAILED DESCRIPTION:
In the present study, a comparison of postoperative pain management in patients who underwent laparoscopic hysterectomy was conducted. The findings indicated that the initial postoperative administration of analgesics occurred later in patients who received peritoneal local anesthetics and SHPB compared to the control group. In addition, VAS values at the first and third hours were found to be lower in the peritoneal local anesthetic and SHPB groups than in the control group. Postoperative pain experienced by patients following gynecologic surgery. It has been reported that approximately 75% of patients experience severe pain. Excessive opioid use in postoperative pain management and the potential for additional complications are also possible. One of the alternative methods to reduce postoperative opioid use is intraperitoneal bupivacaine administration.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent laparoscopic hysterectomy-with or without oophorectomy-
* ASA physical status I-II patients

Exclusion Criteria:

* women with known bupivacaine allergy, anxiety-depressive disorders, fibromyalgia, coagulopathy, eclampsia/preeclampsia, or those who were pregnant were also excluded.
* if they were younger than 18 or older than 65
* underwent epidural catheterisation and/or received additional pain management modalities
* prescribed preoperative antidepressants or gabapentinoids

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprised patients who underwent laparoscopic hysterectomy-with or without oophorectomy-for benign indications (such as myoma uteri, dysfunctional uterine bleeding, uterine prolapse, or precancerous cervical lesions) between July 2024 and December 2024, and who were classified as ASA physical status I-II. Patients were excluded if they were younger than 18 or older than 65, underwent epidural catheterisation and/or received additional pain management modalities (e.g., transversus abdominis plane block, local wound infiltration, quadratus lumborum block), had surgery for malignancy, underwent a different surgical approach (e.g., transvaginal natural orifice transluminal endoscopic surgery), or were prescribed preoperative antidepressants or gabapentinoids.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
VAS (vısual analog scale) | 24 HOUR
  For patients with no pain, VAS was recorded as 0 (zero), and for those with unbearable pain, VAS was recorded as 10 (ten).

CONTACTS AND LOCATIONS:
Locations (1):
- Mardin Artuklu University, Mardin, Turkey (Türkiye)